CLINICAL TRIAL: NCT03143309
Title: WhatsApp Physical Activity Intervention to Promote Walking Among Female University Students in Al-Qassim, Saudi Arabia: A Randomized Controlled Trial.
Brief Title: Physical Activity Intervention to Promote Walking Among Female University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Abdulrahman Al-Mohaimeed, Associate Professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QassimU
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking + WhatsApp (Experimental): The participants assigned to the intervention group will be given a brief (15-minute) orientation where they learn about the importance of exercise, diet, and the benefits of weight reduction. They will be given further instruction on the regular use of the pedometer. They will be enrolled into a WhatsApp group. They will receive 2-3 health-promotional (walking and diet) messages per week via WhatsApp.
  Interventions: Behavioral: Intervention
- WhatsApp Only (Active Comparator): The control participants will be enrolled into a WhatsApp group. They will receive 2-3 non-health related messages per week via WhatsApp.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention — Brief introductory session, pedometer instruction, daily pedometer use, and health messages delivered via WhatsApp 2-3 times per week.
  Other Names: Walking group
  Arms: Walking + WhatsApp
Other: Control — Non-health related messages delivered via WhatsApp 2-3 times per week.
  Other Names: Attention Control
  Arms: WhatsApp Only

SUMMARY:
This study is a parallel group randomized controlled trial among female university students designed to test the effect of a physical activity intervention on daily walking. Both groups will receive messages 2-3 times per week via WhatsApp. Intervention group will receive orientation and wear a pedometer for the study period. The follow-up duration is 3 months.

DETAILED DESCRIPTION:
Background: Sedentary lifestyle is a major risk factor for chronic diseases. The majority of Saudi females do not meet a recommended level of physical activity.

Study Objective: To test the effect of a physical activity intervention on daily walking.

Study Design: Parallel group randomized controlled design among female university students.

Methods: Students will be randomly assigned to either the intervention or the control arm. WhatsApp groups (2 per arm) will be formed within each study arm for communications. The intervention participants will receive a brief (15-minute) orientation on diet, exercise, and benefits of keeping a healthy weight; each will be instructed to wear a pedometer every day for 12-weeks with a daily step goal of 8,000. They will receive 2-3 health-promotional (walking and diet) messages per week via WhatsApp; group interaction is optional. The control group participants will receive 2-3 non-health related messages per week. Average daily steps will be assessed in all participants at baseline and 3-month follow-up using a 7-day pedometer measurement.

ELIGIBILITY:
Inclusion Criteria:

* female
* student enrolled at Qassim University during 2016-2017 academic year
* owns smartphone with internet access
* willing to complete all study requirements

Exclusion Criteria:

* Physical disability that precludes physical activity
* Morbidly obese (Body Mass Index >45 kg/m2)
* Physician recommendation not to exercise

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Walking | Baseline to 3-month follow-up
  Change in 7-day average steps. Measurement tool = Omron pedometer HJ-320

SECONDARY OUTCOMES:
Self-reported walking | Baseline to 3-month follow-up
  Change between baseline and follow-up for walking minutes per week. Measurement tool = International Physical Activity Questionnaire (IPAQ)
Body Mass Index | Baseline to 3-month follow-up
  Change in BMI score between baseline and follow-up. Objective measurement of height and weight.
Barriers to weight management | Baseline to 3-month follow-up
  Change in number of barriers between baseline and follow-up. Measurement tool = Validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Juliann Saquib, PhD, Study Director — College of Medicine, Qassim University
Locations (1):
- Qassim University, Buraidah, Al-Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No